CLINICAL TRIAL: NCT06753786
Title: Early or Delayed Initiation of Venous Thromboembolism Prophylaxis with Heparin in Patients with Hypertensive Intracerebral Hemorrhage
Brief Title: Timing of Venous Thromboembolism Prophylaxis in Patients with Hypertensive Intracerebral Hemorrhage
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pirogov Russian National Research Medical University (Other)
Responsible Party: Principal Investigator, Pryamikov Aleksandr, MD, PhD (DMedSc [Russia]), Associate Professor, Pirogov Russian National Research Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24421102024
Record Dates: First submitted 2024-12-09; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Venous Thromboembolism; Pulmonary Embolism; Intracerebral Hemorrhage; Deep Vein Thrombosis
Keywords: Prophylaxis; Deep vein thrombosis; Pulmonary embolism; Venous thromboembolism; Intracerebral hemorrhage; Anticoagulation; Low molecular weight heparin; Unfractionated heparin
MeSH Terms: conditions — Venous Thromboembolism; Pulmonary Embolism; Cerebral Hemorrhage; Venous Thrombosis | interventions — Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early beginning of venous thromboembolism prophylaxis in patients with intracerebral hemorrhage (Experimental): Participants will receive prophylactic doses of unfractionated heparin or low molecular weight heparin starting within the first 2 days but not earlier than 12 hours after the hospital admission. If a participant is diagnosed with venous thromboembolism after the initiation of venous thromboembolism prophylaxis with heparin, the participant might receive therapeutic doses of unfractionated heparin or low molecular weight heparin by the joint decision of neuroemergency specialist, neurologist, neurosurgeon and vascular surgeon.
  Interventions: Drug: Venous thromboembolism prophylaxis with unfractionated heparin or low molecular weight heparin starting within the first 2 days but not earlier than 12 hours after a hospital admission.
- Delayed beginning of venous thromboembolism prophylaxis in patients with intracerebral hemorrhage (Experimental): Participants will receive prophylactic doses of unfractionated heparin or low molecular weight heparin starting on the 3rd day after the hospital admission. If a participant is diagnosed with venous thromboembolism after the initiation of venous thromboembolism prophylaxis with heparin, the participant might receive therapeutic doses of unfractionated heparin or low molecular weight heparin by the joint decision of neuroemergency specialist, neurologist, neurosurgeon and vascular surgeon.
  Interventions: Drug: Venous thromboembolism prophylaxis with unfractionated heparin or low molecular weight heparin starting on the 3rd day after a hospital admission.

INTERVENTIONS:
Drug: Venous thromboembolism prophylaxis with unfractionated heparin or low molecular weight heparin starting within the first 2 days but not earlier than 12 hours after a hospital admission. — Prophylactic dosage and administration of unfractionated heparin or low molecular weight heparin according to their official prescribing information.
  Arms: Early beginning of venous thromboembolism prophylaxis in patients with intracerebral hemorrhage
Drug: Venous thromboembolism prophylaxis with unfractionated heparin or low molecular weight heparin starting on the 3rd day after a hospital admission. — Prophylactic dosage and administration of unfractionated heparin or low molecular weight heparin according to their official prescribing information.
  Arms: Delayed beginning of venous thromboembolism prophylaxis in patients with intracerebral hemorrhage

SUMMARY:
The objective of this randomized clinical trial is to evaluate the safety and efficiency of different anticoagulation schemes with heparin for venous thromboembolism prevention in patients with hypertensive intracerebral hemorrhage. The main questions it aims to answer are:

* What is the optimal time for the beginning of anticoagulation with heparin to efficiently prevent venous thromboembolism in patients with hypertensive intracerebral hemorrhage? Early beginning (within the first 2 days but not earlier than 12 hours after the admission of a patient) or delayed beginning (on the third day after the admission of a patient)?
* Which of the two timeframes (early or delayed) for anticoagulation beginning is the most safe in terms of bleeding complications including intracerebral hemorrhage expansion?

Researchers will compare the results of early and delayed start of anticoagulation using heparin in patients with hypertensive intracerebral hemorrhage to define the optimal start time for anticoagulation that provides the most favourable efficiency/safety profile.

Participants will:

* Undergo a computed tomography (CT) scan of the brain on hospital admission and then 12-24 hours after the hospital admission and 24 hours after the beginning of venous thromboembolism prophylaxis using heparin;
* Undergo the ultrasound examination of lower extremity deep veins on hospital admission and then once every 7 days;
* Receive prophylactic doses of low molecular weight heparin or unfractionated heparin either beginning within the first 2 days but not earlier than 12 hours after the hospital admission or starting on the 3rd day after the hospital admission.

ELIGIBILITY:
Inclusion Criteria:

* the presence of hypertensive intracerebral hemorrhage

Exclusion Criteria:

* Intracerebral hemorrhage expansion detected on the basis of a computed tomography scan of the brain 12-24 hours after a hospital admission (i.e. before the initiation of venous thromboembolism prophylaxis with heparin)
* Being on an anticoagulant during preadmission period and on day of hospital admission
* Death within the first 2 days after hospital admission
* Detection of venous thromboembolism in a patient at the moment of hospital admission
* Surgical management of hypertensive intracerebral hemorrhage before the beginning of venous thromboembolism prophylaxis using heparin
* The presence of a malignancy (cancer) in a patient at the moment of hospital admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with acute venous thrombosis established using ultrasound examination | From the beginning of venous thromboembolism prophylaxis using heparin until the date of acute venous thrombosis detection or the date of death from any cause, whichever came first, assessed up to hospital discharge but not longer than 6 months.
  Acute venous thrombosis in the study is defined as the development of a blood clot in lower extremity veins and/or pelvic veins and/or inferior vena cava (IVC) and/or IVC tributaries.
Number of participants with pulmonary embolism established using CT pulmonary angiogram | From the beginning of venous thromboembolism prophylaxis using heparin until the date of pulmonary embolism detection or the date of death from any cause, whichever came first, assessed up to hospital discharge but not longer than 6 months.
  Pulmonary embolism in the study is defined as the development of acute fatal or nonfatal pulmonary embolism.
Number of participants with intracerebral hemorrhage expansion detected using brain CT scan | From the beginning of venous thromboembolism prophylaxis using heparin until the date of first documented hemorrhage expansion or the date of death from any cause, whichever came first, assessed up to hospital discharge but not longer than 6 months.
  Intracerebral hemorrhage expansion in the study is defined as hematoma volume absolute increase of > 6 ml and/or relative increase of > 33% compared to its baseline volume.
Number of participants with intracranial bleeding complications requiring urgent neurosurgical management | From the beginning of venous thromboembolism prophylaxis using heparin until the date when the event of interest happens or the date of death from any cause, whichever came first, assessed up to hospital discharge but not longer than 6 months.
Number of participants with clinically significant bleeding beyond the braincase requiring the discontinuation of heparin administration | From the beginning of venous thromboembolism prophylaxis using heparin until the date when the outcome of interest happens or the date of death from any cause, whichever came first, assessed up to hospital discharge but not longer than 6 months.
  Bleeding beyond the braincase (e.g., nosebleed, gastrointestinal bleeding, hemoptysis, etc.) is defined as clinically significant if it: 1) requires transfusion of red blood cells, 2) prolongs a hospitalization, with bleeding as the principal reason, 3) requires surgery to stop the bleeding, or 4) results in death.
Inpatient death rate (mortality) | Starting on the 3rd day after hospital admission until the date of inpatient death or the date of hospital discharge, whichever came first, assessed up to 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Moscow City Clinical Hospital named after V.M. Buyanov, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No